CLINICAL TRIAL: NCT04326296
Title: The Safety, Tolerability and Preliminary Efficacy of PD-L1 Monoclonal Antibody Combined With Lenalidomide in Third-line Post-Treatment of Patients With Microsatellite Stable Advanced Colorectal Cancer: A Phase I Clinical Study
Brief Title: The Safety and Tolerability of PD-L1 Monoclonal Antibody Plus Lenalidomide in The Treatment of Colorectal Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: LiNing (Other Government)
Responsible Party: Sponsor-Investigator, LiNing, Chief Physician, Henan Cancer Hospital
Organization: Henan Cancer Hospital (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRC202001
Record Dates: First submitted 2020-03-26; First posted 2020-03-30 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Experimental): PD-L1 Monoclonal Antibody Combined With Lenalidomide
  Interventions: Drug: PD-L1 Monoclonal Antibody Combined With Lenalidomide

INTERVENTIONS:
Drug: PD-L1 Monoclonal Antibody Combined With Lenalidomide — PD-L1 monoclonal antibody was administered by intravenous drip every 3 weeks.Lenalidomide was administered orally, 25mg once a day on days 1-21 of each repeat cycle of 28 days.

SUMMARY:
This study proposed by increasing dosage and expand the "3 + 3" queue, main component is divided into two phases, phase 1 for dose escalation, according to preliminary data recommended doses starting dose of climbing, the purpose is to evaluate the safety of combination therapy, tolerance, and explore the maximum tolerated dose (MTD) and right dose recommended development stage;Phase 2 was the expansion phase. Patients were included in the expansion study according to the appropriate dose recommended in phase 1, to further evaluate the safety and tolerability of combination therapy, recommend appropriate dose for phase II clinical trial, and preliminarily explore the efficacy of combination therapy.

DETAILED DESCRIPTION:
1. Phase 1 was the dose increasing phase, which was divided into three queues (A, B and C). Each team was included in the group of three people.Cohort B: pd-l1 monoclonal antibody 900mg q3w+ lenalidomide 25mg/d, administration for 21 days/discontinuation for 7 days;Cohort C: pd-l1 monoclonal antibody 20mg/kg q3w+ lenalidomide 25mg/d, administration for 21 days/discontinuation for 7 days.If none of the 3 patients in cohort A in phase 1 showed dose limited toxicity (DLT) within 21 days of their first use, they were enrolled in cohort B, and so on.If 1 of the first 3 subjects in a dose group developed DLT during the DLT observation period after the first combination administration, an additional 3 subjects were added to the dose group.If none of the additional 3 subjects developed DLT, the next incremental dose group was entered.If DLT appears in 1 or more of the additional 3 subjects, the investigator shall decide whether to adjust the regimen, or increase the regimen, or terminate the climb.If DLT appears in 2 or more subjects in the initial 3 subjects of a dose group during the observation period of the first combined DLT, the investigator shall decide whether to adjust the dosing regimen, or increase the dosing regimen, or terminate the climbing.
2. In phase 2, 24 patients will be further included under the initially determined dose level and the appropriate administration regimen. Disease control rate (DCR) will be calculated according to the data obtained in phase 1, and the group with the highest DCR dose will be selected for the expansion study.

ELIGIBILITY:
Inclusion Criteria:

1. Aigned informed consent
2. Only patients aged 18-75 years were enrolled
3. Patients with advanced colorectal cancer diagnosed by pathology and imaging.Note: the presence of distant metastases should be confirmed by a CT or MR scan.Bone scan should be performed if bone metastases are suspected.Local radiotherapy for pain relief is permitted for bone metastases.
4. Measurable lesions based on Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 must be present.Local radiotherapy of target lesions is not allowed.
5. pMMR/MSS advanced colorectal cancer patients with disease progression or intolerance to third-line treatment after failure of current standard third-line treatment
6. ECOG 1 minute or less
7. Tumor specimens that can be used to detect the status of pd-l1, MSI, b-raf and k-ras can be provided.This test requires the patient to provide paraffin embedded biopsy specimens or white slices.
8. White blood cells ≥ 4×109/L, platelets ≥ 100×109/L without transfusion, neutrophil absolute value (ANC) ≥ 1.5×109/L without treatment with granulocyte stimulating factor, and hemoglobin ≥ 90 g/L.
9. Bilirubin ≤ 1.5 times of the upper limit of normal value, and cereal grass and cereal propyl transaminase ≤ 2.5 times of the upper limit of normal value.
10. Serum creatinine ≤ 1.5 times the upper limit of normal value, or GFR>45 ml/min
11. Serum albumin ≥ 25 g/L (2.5g /dL)
12. INR or APTT ≤ 1.5 times ULN
13. Hepatitis B/C surface antigen positive patients need to be tested for Hepatitis B /C virus DNA quantitative test, only < the upper limit of the normal detection value can be included in the group, and long-term use of anti-hb/hc drugs
14. Drug elution time: 28 days or 5 half-lives from the last drug application.

Exclusion Criteria:

1. Allergy to any experimental drug or its excipients, or history of severe allergy, or contraindication to the experimental drug
2. Having a history of autoimmune disease or being active
3. Previous allogeneic bone marrow transplantation or organ transplantation
4. Congenital pulmonary fibrosis, drug-induced pneumonia, organized pneumonia, or ct-confirmed active pneumonia
5. HIV positive
6. Active Hepatitis B /C(Hepatitis B /C viruses have higher quantification than normal)
7. Active stage tuberculosis
8. Uncontrolled cancer pain
9. A live attenuated vaccine was injected within 4 weeks before the study began, or a live attenuated vaccine is expected to be injected during the trial or within 5 months after the end of the trial
10. Previous use of immunotherapy, including CTLA4, anti-PD-1, or anti-PD-L1 monoclonal antibody
11. CT indicates lung active inflammation
12. Systemic administration of glucocorticoids or immunosuppressants within 2 weeks prior to the trial.Inhaled corticosteroids and halocorticoids are allowed
13. Use of hormones is contraindicated
14. Serious cardiovascular disease, myocardial infection, arteriovenous thrombosis or cerebrovascular accident, arrhythmia, unstable angina pectoris within 3 months before the trial
15. Uncontrollable increase in blood pressure or blood sugar
16. History of other malignancies 5 years ago, except for carcinoma in situ of the cervix, non-melanoma skin cancer or stage I uterine cancer
17. Peripheral neuropathy of grade 2 ≥ NCI CTCAE
18. Serum albumin less than 2.5g /dL
19. Uncontrolled or symptomatic hypercalcemia
20. Infection requiring antibiotics within 14 days prior to trial
21. Chronic enteritis
22. Clinically significant active gastrointestinal bleeding
23. Non-diagnostic surgery within 4 weeks before the trial
24. Any other disease for which there is evidence that the use of the experimental drug needs to be restricted
25. Participate in other trials within 30 days prior to the trial or plan to participate in other trials during the trial
26. Receive other experimental drugs within 28 days before the start of the trial
27. Women who are pregnant or lactating, or who plan to become pregnant within 5 months after the end of treatment.Women of childbearing age should undergo a blood pregnancy test 7 days before the start of the trial
28. Use of PD-L1 monoclonal antibody or lenalidomide contraindications
29. MSI-H/dMMR in patients with advanced colorectal cancer

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2020-05-30 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Disease control rate | 1 years
  It is defined as the proportion of complete response, partial response and stable disease
Safety, Tolerability | 1.5 years
  The incidence of serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Ning Li, PhD, Principal Investigator — Henan Cancer Hospital; Suxia Luo, PhD, Principal Investigator — Henan Cancer Hospital
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China